CLINICAL TRIAL: NCT03486457
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY OF THE EFFICACY AND SAFETY OF TOFACITINIB (CP-690,550) IN CHINESE SUBJECTS WITH ACTIVE PSORIATIC ARTHRITIS AND AN INADEQUATE RESPONSE TO AT LEAST ONE CONVENTIONAL SYNTHETIC DMARD
Brief Title: Efficacy And Safety Of Tofacitinib In Chinese Subjects With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921234
Record Dates: First submitted 2018-03-05; First posted 2018-04-03 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-06

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis; tofacitinib; China
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence A (Experimental): Tofacitinib 5 mg BID for 6 months
  Interventions: Drug: Tofacitinib
- Treatment Sequence B (Placebo Comparator): Placebo for 3 months then tofacitinib 5 mg BID for 3 months
  Interventions: Other: Placebo; Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — tablets, 5 mg BID x 6 months
  Arms: Treatment Sequence A
Other: Placebo — tablets, to match tofacitinib 5 mg BID x 3 months
  Arms: Treatment Sequence B
Drug: Tofacitinib — tablets, 5 mg BID x 3 months
  Arms: Treatment Sequence B

SUMMARY:
This is a 6 month study investigating the effectiveness and safety of tofacitinib in treating signs and symptoms and improving physical function in Chinese patients with active psoriatic arthritis and had inadequate response to a conventional synthetic disease modifying anti-rheumatic drug. This is a China alone study.

ELIGIBILITY:
Inclusion Criteria:

* Chinese patients
* Active arthritis at screening/baseline as indicated by >/= 3 tender/painful and 3 swollen joints
* Active plaque psoriasis at screening
* Inadequate response to at least one conventional synthetic DMARD

Exclusion Criteria:

* Non-plaque forms of psoriasis (with exception of nail psoriasis)
* History of autoimmune rheumatic disease other than PsA; also prior history of or current, rheumatic inflammatory disease other than PsA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- China (38):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University/Rheumatology Department, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Army Medical University, PLA, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - The Third Hospital of Hebei Medical University, Rheumatology and Immunology Department, Shijiazhuang, Hebei
  - Rheumatology Department, The first Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Department of Rheumatology, The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Department of Rheumatology ,The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Department of Rheumatology, Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiu Jiang No.1 People's Hospital, Jiujiang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First hospital of Jilin University, Changchun, Jilin
  - Linyi People's Hospital, Linyi, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Department of Rheumatology and Immunology,West China Hospital，Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Rheumatology and Immunology Department, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Rheumatology and Immunology Department, Xuanwu Hospital Capital Medical University, Beijing
  - Huashan Hospital, Fudan University, Shanghai
  - Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Gladman DD, Dougados M, Marzo-Ortega H, Cadatal MJ, Agarwal E, Kinch CD, Nash P. Long-term tofacitinib efficacy and safety in psoriatic arthritis with or without prior biologic DMARD exposure: a post hoc analysis. Rheumatol Adv Pract. 2025 Jan 21;9(2):rkaf008. doi: 10.1093/rap/rkaf008. eCollection 2025. PMID 40241921
- [Derived] Leng X, Lin W, Liu S, Kanik K, Wang C, Wan W, Jiang Z, Liu Y, Liu S, Zhang Z, Zhang Z, Xu J, Tan W, Hu J, Li J, Liu J, Gunay LM, Dina O, Kinch C, Zeng X. Efficacy and safety of tofacitinib in Chinese patients with active psoriatic arthritis: a phase 3, randomised, double-blind, placebo-controlled study. RMD Open. 2023 Jan;9(1):e002559. doi: 10.1136/rmdopen-2022-002559. PMID 36720560
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921234

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three hundred and forty five participants were screened and a total of 204 participants assigned to study treatment were treated (136 in the tofacitinib 5 mg BID group and 68 in the placebo → tofacitinib 5 mg twice a day [BID] group). Safety data was planned to be collected and reported for both: from Baseline to Month 3 and from Baseline to Month 6.
Groups:
- Tofacitinib: Participants received Tofacitinib 5 milligram (mg) twice daily (BID) for 6 months.
- Placebo Then Tofacitinib: Participants received tofacitinib matching placebo tablets BID for 3 months, followed by tofacitinib tablets 5 mg BID for next 3 months (up to Month 6).
Period: Up to Month 3
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Started | 136 | 68
Completed | 129 | 63
Not Completed | 7 | 5
Not completed — Adverse Event | 2 | 5
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Failure to Meet Randomization Criteria | 2 | 0
Not completed — Other | 1 | 0
Period: Month 3 to Month 6
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Started | 129 | 63
Completed | 126 | 61
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: included all participants who received at least one dose of the study drug (tofacitinib or placebo)
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib | Placebo Then Tofacitinib | Total
Number analyzed (Participants) | 136 | 68 | 204
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.3 (11.59) | 43.9 (10.40) | 44.8 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 26 | 83
  Male | 79 | 42 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 136 | 68 | 204
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 136 | 68 | 204
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Month 3
Description: ACR50 response: greater than or equal to (≥) 50% improvement in tender (TJC) and swollen joint counts (SJC) and ≥50% improvement in 3 of the 5 remaining ACR-core set measures: patient (PtGA) and physician global assessments (PhyGA), pain, disability (Health Assessment Questionnaire - Disability Index [HAQ-DI], scored from 0 to 3), and an acute-phase reactant (C-reactive protein [CRP]). TJC was based on 68 joints and SJC was based on 66 joints. PtGA, PhyGA and Pain were VAS on a scale of 0-100 millimeter (mm).
Time Frame: Month 3
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Missing response (MR) was considered to be non-response (NR) (MR=NR).
Measure: Number; unit: Percentage of participants
Groups:
- Tofacitinib: Participants received Tofacitinib 5 mg BID for 6 months.
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 136 | 68
Percentage of participants | 38.24 | 5.88
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; The normal approximation to the difference in binomial proportions was used to test the difference between tofacitinib 5 mg BID and placebo and to generate 95% CI and p-value for the difference in response rates; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 32.35, 95% CI 2-sided [22.45 to 42.25], Standard Error of Mean 5.05

2. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 2, Month 1, 2, 3, 4, and 6
Description: ACR20 response:≥20% improvement in TJC and SJC and ≥20% improvement in 3 of the 5 remaining ACR-core set measures: PtGA and PhyGA, pain, disability (HAQ-DI, scored from 0 to 3), and a CRP. TJC was based on 68 joints and SJC was based on 66 joints. PtGA, PhyGA and Pain were VAS on a scale of 0-100 mm.
Time Frame: Week 2, Month 1, 2, 3, 4, and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  MR was considered to be NR (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 136 | 68
Percentage of participants
  Week 2 | 22.79 | 7.35
  Month 1 | 38.97 | 8.82
  Month 2 | 61.76 | 10.29
  Month 3 | 64.71 | 27.94
  Month 4 | 69.85 | 45.59
  Month 6 | 72.79 | 58.82
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 2: The normal approximation to the difference in binomial proportions was used to test the difference between the two treatment arms and to generate 95% CI and p-value for the difference in response rates; Test type: Superiority; p = 0.0013, Normal approximation; Difference in percentage of participants = 15.44, 95% CI 2-sided [6.05 to 24.83], Standard Error of Mean 4.79
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1: The normal approximation to the difference in binomial proportions was used to test the difference between the two treatment arms and to generate 95% CI and p-value for the difference in response rates; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 30.15, 95% CI 2-sided [19.53 to 40.76], Standard Error of Mean 5.41
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 2: The normal approximation to the difference in binomial proportions was used to test the difference between the two treatment arms and to generate 95% CI and p-value for the difference in response rates; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 51.47, 95% CI 2-sided [40.57 to 62.37], Standard Error of Mean 5.56
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3: The normal approximation to the difference in binomial proportions was used to test the difference between the two treatment arms and to generate 95% CI and p-value for the difference in response rates; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 36.76, 95% CI 2-sided [23.41 to 50.12], Standard Error of Mean 6.81
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 4: The normal approximation to the difference in binomial proportions was used to test the difference between the two treatment arms and to generate 95% CI and p-value for the difference in response rates; Test type: Superiority; p = 0.0008, Normal approximation; Difference in percentage of participants = 24.26, 95% CI 2-sided [10.14 to 38.39], Standard Error of Mean 7.21
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6: The normal approximation to the difference in binomial proportions was used to test the difference between the two treatment arms and to generate 95% CI and p-value for the difference in response rates; Test type: Superiority; p = 0.0486, Normal approximation; Difference in percentage of participants = 13.97, 95% CI 2-sided [0.09 to 27.85], Standard Error of Mean 7.08

3. Secondary Outcome: Percentage of Participants Achieving ACR70 Response at Week 2, Month 1, 2, 3, 4, and 6
Description: ACR70 response:≥70% improvement in TJC and SJC and ≥70% improvement in 3 of the 5 remaining ACR-core set measures: PtGA and PhyGA, pain, disability (HAQ-DI, scored from 0 to 3), and a CRP. TJC was based on 68 joints and SJC was based on 66 joints. PtGA, PhyGA and Pain were VAS on a scale of 0-100 mm.
Time Frame: Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 136 | 68
Percentage of participants
  Week 2 | 1.47 | 0
  Month 1 | 2.21 | 0
  Month 2 | 8.82 | 1.47
  Month 3 | 14.71 | 1.47
  Month 4 | 20.59 | 7.35
  Month 6 | 36.76 | 23.53
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4730, Normal approximation; Difference in percentage of participants = 1.10, 95% CI 2-sided [-1.90 to 4.10], Standard Error of Mean 1.53
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.2792, Normal approximation; Difference in percentage of participants = 1.83, 95% CI 2-sided [-1.48 to 5.14], Standard Error of Mean 1.69
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.0095, Normal approximation; Difference in percentage of participants = 7.35, 95% CI 2-sided [1.79 to 12.91], Standard Error of Mean 2.84
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 13.24, 95% CI 2-sided [6.63 to 19.84], Standard Error of Mean 3.37
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.0048, Normal approximation; Difference in percentage of participants = 13.24, 95% CI 2-sided [4.03 to 22.44], Standard Error of Mean 4.69
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.0449, Normal approximation; Difference in percentage of participants = 13.24, 95% CI 2-sided [0.30 to 26.17], Standard Error of Mean 6.60

4. Secondary Outcome: Percentage of Participants Achieving ACR50 Response at Week 2, Month 1, 2, 4, and 6
Description: ACR50 response:≥50% improvement in TJC and SJC and ≥50% improvement in 3 of the 5 remaining ACR-core set measures: PtGA and PhyGA, pain, disability (HAQ-DI, scored from 0 to 3), and a CRP. TJC was based on 68 joints and SJC was based on 66 joints. PtGA, PhyGA and Pain were VAS on a scale of 0-100 mm.
Time Frame: Week 2, Month 1, 2, 4, and 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 136 | 68
Percentage of participants
  Week 2 | 4.41 | 1.47
  Month 1 | 9.56 | 1.47
  Month 2 | 30.15 | 2.94
  Month 4 | 41.18 | 19.12
  Month 6 | 55.15 | 36.76
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1985, Normal approximation; Difference in percentage of participants = 2.94, 95% CI 2-sided [-1.54 to 7.42], Standard Error of Mean 2.29
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0055, Normal approximation; Difference in percentage of participants = 8.09, 95% CI 2-sided [2.38 to 13.80], Standard Error of Mean 2.91
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 27.21, 95% CI 2-sided [18.51 to 35.90], Standard Error of Mean 4.44
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.0005, Normal approximation; Difference in percentage of participants = 22.06, 95% CI 2-sided [9.58 to 34.54], Standard Error of Mean 6.37
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.0111, Normal approximation; Difference in percentage of participants = 18.38, 95% CI 2-sided [4.20 to 32.57], Standard Error of Mean 7.24

5. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 2, Month 1, 2, 3, 4, and 6
Description: The HAQ-DI assessed the degree of difficulty a participant had experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consisted of 2-3 items. For each question in the questionnaire, the level of difficulty was scored from 0 to 3 with 0 representing "no difficulty," 1 as "some difficulty," 2 as "much difficulty," and 3 as "unable to do". The HAQ-DI score was the average of the non-missing domain scores. If >2 domain scores were missing, HAQ-DI score was considered missing. A higher score represented a more limited physical functional status/ability.
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4, and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Here "Number of Participants Analyzed" indicates participants included in the MMRM.
  Here "Number analyzed" signifies participants evaluable for this OM at the specific visit.
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 135 | 67
unit on a scale
  Week 2: number analyzed (Participants) | 134 | 67
  Week 2 | -0.14 (0.025) | -0.03 (0.036)
  Month 1: number analyzed (Participants) | 133 | 64
  Month 1 | -0.18 (0.026) | -0.05 (0.037)
  Month 2: number analyzed (Participants) | 125 | 64
  Month 2 | -0.28 (0.028) | -0.07 (0.039)
  Month 3: number analyzed (Participants) | 127 | 62
  Month 3 | -0.30 (0.031) | -0.08 (0.044)
  Month 4: number analyzed (Participants) | 129 | 62
  Month 4 | -0.32 (0.026) | -0.23 (0.038)
  Month 6: number analyzed (Participants) | 126 | 61
  Month 6 | -0.38 (0.025) | -0.31 (0.036)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 2: Analysis performed using mixed model for repeated measures (MMRM) which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0097, Mixed Models Analysis; LS mean difference = -0.11, 95% CI 2-sided [-0.20 to -0.03], Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0043, Mixed Models Analysis; LS mean difference = -0.13, 95% CI 2-sided [-0.22 to -0.04], Standard Error of Mean 0.045
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 2: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.21, 95% CI 2-sided [-0.30 to -0.11], Standard Error of Mean 0.048
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.22, 95% CI 2-sided [-0.32 to -0.11], Standard Error of Mean 0.053
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 4: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0535, Mixed Models Analysis; LS mean difference = -0.09, 95% CI 2-sided [-0.18 to 0.00], Standard Error of Mean 0.046
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0940, Mixed Models Analysis; LS mean difference = -0.07, 95% CI 2-sided [-0.16 to 0.01], Standard Error of Mean 0.044

6. Secondary Outcome: HAQ-DI Response (Decrease From Baseline ≥0.30) Rate for Participants With Baseline HAQ-DI ≥0.30 at Week 2, Month 1, 2, 3, 4, and 6
Description: Rate was measured in terms of percentage of participants with HAQ-DI response. The HAQ-DI assessed the degree of difficulty a participant had experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consisted of 2-3 items. For each question in the questionnaire, the level of difficulty was scored from 0 to 3 with 0 representing "no difficulty," 1 as "some difficulty," 2 as "much difficulty," and 3 as "unable to do". The HAQ-DI score was the average of the non-missing domain scores. If >2 domain scores were missing, HAQ-DI score was considered missing. A higher score represented a more limited physical functional status/ability.
Time Frame: Week 2, Month 1, 2, 3, 4, and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline HAQ-DI ≥0.30. MR was considered to be NR (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 83 | 39
Percentage of participants
  Week 2 | 36.14 | 23.08
  Month 1 | 37.35 | 33.33
  Month 2 | 60.24 | 38.46
  Month 3 | 65.06 | 41.03
  Month 4 | 63.86 | 51.28
  Month 6 | 73.49 | 66.67
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1270, Normal approximation; Difference in percentage of participants = 13.07, 95% CI 2-sided [-3.72 to 29.85], Standard Error of Mean 8.56
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.6634, Normal approximation; Difference in percentage of participants = 4.02, 95% CI 2-sided [-14.07 to 22.10], Standard Error of Mean 9.23
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.0214, Normal approximation; Difference in percentage of participants = 21.78, 95% CI 2-sided [3.23 to 40.33], Standard Error of Mean 9.46
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.0110, Normal approximation; Difference in percentage of participants = 24.03, 95% CI 2-sided [5.50 to 42.57], Standard Error of Mean 9.46
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.1896, Normal approximation; Difference in percentage of participants = 12.57, 95% CI 2-sided [-6.21 to 31.36], Standard Error of Mean 9.58
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.4466, Normal approximation; Difference in percentage of participants = 6.83, 95% CI 2-sided [-10.75 to 24.41], Standard Error of Mean 8.97

7. Secondary Outcome: HAQ-DI Response (Decrease From Baseline ≥0.35) Rate for Participants With Baseline HAQ-DI ≥0.35 at Week 2, Month 1, 2, 3, 4, and 6
Description: as for outcome 6
Time Frame: Week 2, Month 1, 2, 3, 4, and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline HAQ-DI ≥0.35. MR was considered to be NR (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 83 | 39
Percentage of participants
  Week 2 | 36.14 | 23.08
  Month 1 | 37.35 | 33.33
  Month 2 | 60.24 | 38.46
  Month 3 | 65.06 | 41.03
  Month 4 | 63.86 | 51.28
  Month 6 | 73.49 | 66.67
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1270, Normal approximation; Difference in percentage of participants = 13.07, 95% CI 2-sided [-3.72 to 29.85], Standard Error of Mean 8.56
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.6634, Normal approximation; Difference in percentage of participants = 4.02, 95% CI 2-sided [-14.07 to 22.10], Standard Error of Mean 9.23
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.0214, Normal approximation; Difference in percentage of participants = 21.78, 95% CI 2-sided [3.23 to 40.33], Standard Error of Mean 9.46
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.0110, Normal approximation; Difference in percentage of participants = 24.03, 95% CI 2-sided [5.50 to 42.57], Standard Error of Mean 9.46
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.1896, Normal approximation; Difference in percentage of participants = 12.57, 95% CI 2-sided [-6.21 to 31.36], Standard Error of Mean 9.58
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.4466, Normal approximation; Difference in percentage of participants = 6.83, 95% CI 2-sided [-10.75 to 24.41], Standard Error of Mean 8.97

8. Secondary Outcome: Change From Baseline in Swollen Joint Count at Week 2, Month 1, 2, 3, 4, and 6
Description: Swollen joint count was an assessment on 66 joints (temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeals, thumb interphalangeal, proximal interphalangeals, distal interphalangeals, knee, ankle, tarsus, metatarsophalangeals, great toe interphalangeal, proximal and distal interphalangeals combined). Artificial joints were not assessed. Each joint was assessed for swelling as: Present/Absent/Not Done/Not Applicable (used for artificial or missing joints).
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Joint count
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 135 | 67
Joint count
  Week 2: number analyzed (Participants) | 131 | 67
  Week 2 | -3.04 (0.367) | -0.34 (0.516)
  Month 1: number analyzed (Participants) | 126 | 62
  Month 1 | -4.06 (0.409) | -0.27 (0.582)
  Month 2: number analyzed (Participants) | 117 | 58
  Month 2 | -5.55 (0.437) | -0.66 (0.622)
  Month 3: number analyzed (Participants) | 123 | 60
  Month 3 | -6.42 (0.489) | -0.57 (0.697)
  Month 4: number analyzed (Participants) | 115 | 57
  Month 4 | -7.28 (0.336) | -4.08 (0.476)
  Month 6: number analyzed (Participants) | 115 | 57
  Month 6 | -8.07 (0.386) | -5.48 (0.545)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -2.70, 95% CI 2-sided [-3.95 to -1.45], Standard Error of Mean 0.633
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -3.79, 95% CI 2-sided [-5.20 to -2.39], Standard Error of Mean 0.711
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -4.89, 95% CI 2-sided [-6.39 to -3.39], Standard Error of Mean 0.760
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -5.85, 95% CI 2-sided [-7.53 to -4.17], Standard Error of Mean 0.852
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -3.20, 95% CI 2-sided [-4.35 to -2.04], Standard Error of Mean 0.583
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS mean difference = -2.59, 95% CI 2-sided [-3.91 to -1.27], Standard Error of Mean 0.668

9. Secondary Outcome: Change From Baseline in Tender/Painful Joint Count at Week 2, Month 1, 2, 3, 4, and 6
Description: Tender/painful joint count was an assessment on 68 joints (temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeals, thumb interphalangeal, proximal interphalangeals, distal interphalangeals, hip, knee, ankle, tarsus, metatarsophalangeals, great toe interphalangeal, proximal and distal interphalangeals combined). Artificial joints were not assessed. Each joint was assessed for tenderness/pain as: Present/Absent/Not Done/Not Applicable (used for artificial or missing joints).
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Joint count
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 135 | 67
Joint count
  Week 2: number analyzed (Participants) | 131 | 67
  Week 2 | -3.19 (0.585) | 0.21 (0.825)
  Month 1: number analyzed (Participants) | 126 | 62
  Month 1 | -5.38 (0.589) | -0.35 (0.838)
  Month 2: number analyzed (Participants) | 117 | 58
  Month 2 | -7.44 (0.588) | -1.76 (0.837)
  Month 3: number analyzed (Participants) | 123 | 60
  Month 3 | -8.90 (0.637) | -1.89 (0.910)
  Month 4: number analyzed (Participants) | 115 | 57
  Month 4 | -10.15 (0.617) | -6.19 (0.878)
  Month 6: number analyzed (Participants) | 115 | 57
  Month 6 | -11.91 (0.638) | -9.51 (0.906)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0010, Mixed Models Analysis; LS mean difference = -3.40, 95% CI 2-sided [-5.40 to -1.40], Standard Error of Mean 1.012
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -5.03, 95% CI 2-sided [-7.05 to -3.01], Standard Error of Mean 1.024
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -5.68, 95% CI 2-sided [-7.70 to -3.66], Standard Error of Mean 1.023
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -7.01, 95% CI 2-sided [-9.20 to -4.82], Standard Error of Mean 1.111
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0003, Mixed Models Analysis; LS mean difference = -3.95, 95% CI 2-sided [-6.07 to -1.83], Standard Error of Mean 1.073
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.0323, Mixed Models Analysis; LS mean difference = -2.39, 95% CI 2-sided [-4.58 to -0.20], Standard Error of Mean 1.108

10. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain Visual Analog Scale (VAS) at Week 2, Month 1, 2, 3, 4, and 6
Description: Participants were assessed the severity of their arthritis pain using a 100 mm VAS by placing a mark on the scale between 0 (no pain) and 100 (most severe pain).
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 135 | 67
mm
  Week 2: number analyzed (Participants) | 134 | 67
  Week 2 | -9.7 (1.429) | -3.13 (2.025)
  Month 1: number analyzed (Participants) | 132 | 63
  Month 1 | -14.07 (1.421) | -2.37 (2.038)
  Month 2: number analyzed (Participants) | 125 | 62
  Month 2 | -18.80 (1.606) | -2.66 (2.286)
  Month 3: number analyzed (Participants) | 127 | 62
  Month 3 | -23.07 (1.735) | -1.20 (2.478)
  Month 4: number analyzed (Participants) | 126 | 61
  Month 4 | -24.79 (1.641) | -17.84 (2.346)
  Month 6: number analyzed (Participants) | 124 | 59
  Month 6 | -29.37 (1.692) | -26.27 (2.435)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0087, Mixed Models Analysis; LS mean difference = -6.57, 95% CI 2-sided [-11.46 to -1.68], Standard Error of Mean 2.481
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -11.70, 95% CI 2-sided [-16.60 to -6.79], Standard Error of Mean 2.487
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -16.14, 95% CI 2-sided [-21.66 to -10.63], Standard Error of Mean 2.796
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -21.87, 95% CI 2-sided [-27.84 to -15.90], Standard Error of Mean 3.027
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0163, Mixed Models Analysis; LS mean difference = -6.94, 95% CI 2-sided [-12.60 to -1.29], Standard Error of Mean 2.865
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.2977, Mixed Models Analysis; LS mean difference = -3.10, 95% CI 2-sided [-8.95 to 2.76], Standard Error of Mean 2.967

11. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis (VAS) at Week 2, Month 1, 2, 3, 4, and 6
Description: Participants answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" The participant's response was recorded using a 100 mm VAS by placing a mark on the scale between 0 (Very well) and 100 (Very poorly).
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 135 | 67
mm
  Week 2: number analyzed (Participants) | 134 | 67
  Week 2 | -13.67 (1.521) | -7.52 (2.157)
  Month 1: number analyzed (Participants) | 131 | 63
  Month 1 | -17.89 (1.593) | -4.80 (2.283)
  Month 2: number analyzed (Participants) | 125 | 62
  Month 2 | -22.49 (1.679) | -9.33 (2.392)
  Month 3: number analyzed (Participants) | 127 | 62
  Month 3 | -26.02 (1.825) | -7.25 (2.606)
  Month 4: number analyzed (Participants) | 126 | 60
  Month 4 | -28.68 (1.613) | -21.67 (2.316)
  Month 6: number analyzed (Participants) | 124 | 59
  Month 6 | -33.49 (1.669) | -28.35 (2.404)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0211, Mixed Models Analysis; LS mean difference = -6.15, 95% CI 2-sided [-11.37 to -0.93], Standard Error of Mean 2.646
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -13.08, 95% CI 2-sided [-18.59 to -7.58], Standard Error of Mean 2.790
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -13.16, 95% CI 2-sided [-18.93 to -7.38], Standard Error of Mean 2.928
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -18.77, 95% CI 2-sided [-25.06 to -12.49], Standard Error of Mean 3.187
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0140, Mixed Models Analysis; LS mean difference = -7.01, 95% CI 2-sided [-12.59 to -1.43], Standard Error of Mean 2.827
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.0811, Mixed Models Analysis; LS mean difference = -5.14, 95% CI 2-sided [-10.93 to 0.64], Standard Error of Mean 2.931

12. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis (VAS) at Week 2, Month 1, 2, 3, 4, and 6
Description: The blinded investigator or qualified assessor assessed how the participant's overall arthritis appeared at the time of the visit. This was an evaluation based on the participant's disease signs, functional capacity and physical examination, and should be independent of the Patient's Global Assessment of Arthritis. The investigator's response was recorded using a 100 mm VAS by placing a mark on the scale between 0 (Very good) and 100 (Very poor).
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 135 | 67
mm
  Week 2: number analyzed (Participants) | 131 | 67
  Week 2 | -11.94 (1.126) | -2.30 (1.579)
  Month 1: number analyzed (Participants) | 126 | 62
  Month 1 | -17.10 (1.324) | -7.58 (1.887)
  Month 2: number analyzed (Participants) | 117 | 58
  Month 2 | -25.16 (1.419) | -8.19 (2.024)
  Month 3: number analyzed (Participants) | 123 | 60
  Month 3 | -29.45 (1.436) | -11.03 (2.053)
  Month 4: number analyzed (Participants) | 115 | 58
  Month 4 | -33.33 (1.413) | -26.11 (2.004)
  Month 6: number analyzed (Participants) | 114 | 57
  Month 6 | -38.79 (1.307) | -31.13 (1.851)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -9.64, 95% CI 2-sided [-13.46 to -5.81], Standard Error of Mean 1.939
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -9.52, 95% CI 2-sided [-14.07 to -4.98], Standard Error of Mean 2.305
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -16.97, 95% CI 2-sided [-21.85 to -12.10], Standard Error of Mean 2.472
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -18.42, 95% CI 2-sided [-23.36 to -13.48], Standard Error of Mean 2.506
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0037, Mixed Models Analysis; LS mean difference = -7.22, 95% CI 2-sided [-12.06 to -2.38], Standard Error of Mean 2.453
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.0009, Mixed Models Analysis; LS mean difference = -7.66, 95% CI 2-sided [-12.13 to -3.18], Standard Error of Mean 2.267

13. Secondary Outcome: Change From Baseline in CRP at Week 2, Month 1, 2, 3, 4, and 6
Description: Blood samples were collected at each visit (except follow-up) for analysis of CRP using an assay by the central laboratory. The test for CRP was a laboratory measurement for evaluation of an acute phase reactant of inflammation. A decrease in the level of CRP indicated reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 135 | 67
mg/L
  Week 2: number analyzed (Participants) | 131 | 66
  Week 2 | -8.63 (0.641) | -1.42 (0.904)
  Month 1: number analyzed (Participants) | 126 | 62
  Month 1 | -9.37 (0.673) | -1.50 (0.958)
  Month 2: number analyzed (Participants) | 117 | 58
  Month 2 | -9.24 (0.679) | -1.83 (0.967)
  Month 3: number analyzed (Participants) | 123 | 60
  Month 3 | -9.78 (0.700) | -1.98 (1.001)
  Month 4: number analyzed (Participants) | 115 | 57
  Month 4 | -10.28 (0.354) | -10.58 (0.503)
  Month 6: number analyzed (Participants) | 115 | 56
  Month 6 | -10.24 (0.445) | -8.95 (0.638)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -7.20, 95% CI 2-sided [-9.39 to -5.02], Standard Error of Mean 1.108
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -7.87, 95% CI 2-sided [-10.18 to -5.56], Standard Error of Mean 1.171
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -7.41, 95% CI 2-sided [-9.74 to -5.08], Standard Error of Mean 1.182
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -7.80, 95% CI 2-sided [-10.21 to -5.39], Standard Error of Mean 1.221
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.6264, Mixed Models Analysis; LS mean difference = 0.30, 95% CI 2-sided [-0.91 to 1.51], Standard Error of Mean 0.615
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.1008, Mixed Models Analysis; LS mean difference = -1.29, 95% CI 2-sided [-2.82 to 0.25], Standard Error of Mean 0.778

14. Secondary Outcome: Physician's Global Assessment of Psoriasis (PGA-PsO) Response Rates for Participants With Baseline PGA-PsO ≥2 at Month 1, 3 and 6
Description: PGA-PsO response : PGA-PsO = 0 or 1 and decrease from baseline in PGA-PsO ≥2. Rate was measured in terms of percentage of participants with PGA-PsO response. The PGA-PsO was scored on a 5-point scale, reflecting a global consideration of the erythema, induration and scaling across all psoriatic lesions. Average erythema, induration and scaling were scored separately over the whole body according to a 5-point severity scale, scored as 0 (none), 1, 2, 3, or 4 (most severe). The severity scores were summed and averaged after which the total average was rounded to the nearest whole number score to determine the PGA-PsO score.
Time Frame: Month 1, 3 and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline PGA-PsO ≥2. MR was considered to be NR (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 106 | 51
Percentage of participants
  Month 1 | 0.94 | 0.00
  Month 3 | 9.43 | 1.96
  Month 6 | 10.38 | 21.57
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.8032, Normal approximation; Difference in percentage of participants = 0.44, 95% CI 2-sided [-3.02 to 3.90], Standard Error of Mean 1.77
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.0298, Normal approximation; Difference in percentage of participants = 7.47, 95% CI 2-sided [0.73 to 14.21], Standard Error of Mean 3.44
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.0840, Normal approximation; Difference in percentage of participants = -11.19, 95% CI 2-sided [-23.88 to 1.50], Standard Error of Mean 6.48

15. Secondary Outcome: Change From Baseline in PGA-PsO for Participants With Baseline PGA-PsO>0 at Month 1, 3 and 6
Description: The PGA-PsO was scored on a 5-point scale, reflecting a global consideration of the erythema, induration and scaling across all psoriatic lesions. Average erythema, induration and scaling were scored separately over the whole body according to a 5-point severity scale, scored as 0 (none), 1, 2, 3, or 4 (most severe). The severity scores were summed and averaged after which the total average was rounded to the nearest whole number score to determine the PGA-PsO score.
Time Frame: Baseline, Month 1, 3 and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo). Analysis only included participants in FAS with Baseline PGA-PsO >0.
  Here "Number of Participants Analyzed" indicates participants included in the MMRM.
  Here "Number analyzed" signifies participants evaluable for this OM at the specific visit.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 130 | 63
Unit on a scale
  Month 1: number analyzed (Participants) | 123 | 61
  Month 1 | -0.66 (0.064) | -0.31 (0.091)
  Month 3: number analyzed (Participants) | 119 | 58
  Month 3 | -1.12 (0.080) | -0.52 (0.114)
  Month 6: number analyzed (Participants) | 112 | 54
  Month 6 | -1.25 (0.089) | -1.26 (0.128)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0020, Mixed Models Analysis; LS mean difference = -0.35, 95% CI 2-sided [-0.57 to -0.13], Standard Error of Mean 0.111
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.59, 95% CI 2-sided [-0.87 to -0.32], Standard Error of Mean 0.140
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.9678, Mixed Models Analysis; LS mean difference = 0.01, 95% CI 2-sided [-0.30 to 0.31], Standard Error of Mean 0.156

16. Secondary Outcome: Psoriasis Area and Severity Index (PASI) 75 Response Rates at Month 1, 3 and 6 in Participants With Baseline Psoriatic Body Surface Area (BSA) ≥3% and Baseline PASI >0
Description: PASI75 response: ≥75% improvement from baseline in PASI. Rate was measured in terms of percentage of participants with PASI75 response. PASI quantified the severity of a participant's psoriasis based on both lesion severity and the percent of BSA affected. PASI score ranged from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI was only performed if ≥3% of participant's BSA was affected at baseline.
Time Frame: Month 1, 3 and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline BSA ≥3% and Baseline PASI >0.
  MR was considered to be NR (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 75 | 27
Percentage of participants
  Month 1 | 18.67 | 3.70
  Month 3 | 36.00 | 11.11
  Month 6 | 41.33 | 59.26
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0097, Normal approximation; Difference in percentage of participants = 14.96, 95% CI 2-sided [3.63 to 26.30], Standard Error of Mean 5.78
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.0024, Normal approximation; Difference in percentage of participants = 24.89, 95% CI 2-sided [8.81 to 40.97], Standard Error of Mean 8.20
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.1042, Normal approximation; Difference in percentage of participants = -17.93, 95% CI 2-sided [-39.55 to 3.70], Standard Error of Mean 11.03

17. Secondary Outcome: Percent Change From Baseline in PASI Score at Month 1, 3 and 6 for Participants With Baseline BSA ≥3% and Baseline PASI >0
Description: PASI quantified the severity of a participant's psoriasis based on both lesion severity and the percentage of BSA affected. PASI was a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. PASI score ranged from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI was only performed if ≥3% of participant's BSA was affected at baseline.
Time Frame: Baseline, Month 1, 3 and 6
Population: The unit of Percentage is for percent change from baseline: (change from baseline / baseline value)*100% FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo). Analysis only included participants in FAS with Baseline BSA ≥3% and Baseline PASI >0.
  Here "Number of Participants Analyzed" indicates participants included in the MMRM.
  Here "Number analyzed" signifies participants evaluable for this OM at the specific visit.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 72 | 25
Percentage
  Month 1: number analyzed (Participants) | 70 | 25
  Month 1 | -42.23 (4.021) | -16.34 (6.750)
  Month 3: number analyzed (Participants) | 63 | 24
  Month 3 | -60.86 (4.660) | -25.95 (7.637)
  Month 6: number analyzed (Participants) | 59 | 23
  Month 6 | -62.72 (5.617) | -68.03 (9.065)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0014, Mixed Models Analysis; LS mean difference = -25.89, 95% CI 2-sided [-41.49 to -10.29], Standard Error of Mean 7.858
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS mean difference = -34.91, 95% CI 2-sided [-52.69 to -17.13], Standard Error of Mean 8.948
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.6200, Mixed Models Analysis; LS mean difference = 5.31, 95% CI 2-sided [-15.90 to 26.51], Standard Error of Mean 10.663

18. Secondary Outcome: Percent Change From Baseline in PASI Clinical Component Scores at Month 1, 3 and 6 for Participants With Baseline BSA ≥3% and Baseline PASI >0
Description: PASI quantified the severity of a participant's psoriasis based on both lesion severity and the percentage of BSA affected. PASI was a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. PASI was only performed if ≥3% of participant's BSA was affected at baseline. The PASI clinical component scores (erythema, induration and scaling) range from 0.0 to 24.0, with higher scores representing increasing severity of psoriasis.
Time Frame: Baseline, Month 1, 3 and 6
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 72 | 25
Percentage
  Month 1: Erythema: number analyzed (Participants) | 70 | 25
  Month 1: Erythema | -44.53 (5.553) | -4.89 (9.335)
  Month 1: Induration: number analyzed (Participants) | 70 | 25
  Month 1: Induration | -39.91 (4.329) | -14.73 (7.261)
  Month 1: Scaling: number analyzed (Participants) | 70 | 25
  Month 1: Scaling | -37.25 (5.331) | -15.94 (8.954)
  Month 3: Erythema: number analyzed (Participants) | 63 | 24
  Month 3: Erythema | -63.49 (5.471) | -14.38 (8.993)
  Month 3: Induration: number analyzed (Participants) | 63 | 24
  Month 3: Induration | -58.71 (4.935) | -29.01 (8.082)
  Month 3: Scaling: number analyzed (Participants) | 63 | 24
  Month 3: Scaling | -56.91 (5.575) | -20.13 (9.153)
  Month 6: Erythema: number analyzed (Participants) | 59 | 23
  Month 6: Erythema | -61.40 (5.543) | -68.43 (8.911)
  Month 6: Induration: number analyzed (Participants) | 59 | 23
  Month 6: Induration | -60.47 (6.468) | -69.63 (10.430)
  Month 6: Scaling: number analyzed (Participants) | 59 | 23
  Month 6: Scaling | -63.20 (6.088) | -63.89 (9.803)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Erythema: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0004, Mixed Models Analysis; LS mean difference = -39.65, 95% CI 2-sided [-61.21 to -18.08], Standard Error of Mean 10.862
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Induration: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0037, Mixed Models Analysis; LS mean difference = -25.18, 95% CI 2-sided [-41.97 to -8.40], Standard Error of Mean 8.453
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Scaling: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0438, Mixed Models Analysis; LS mean difference = -21.30, 95% CI 2-sided [-42.00 to -0.61], Standard Error of Mean 10.423
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Erythema: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -49.11, 95% CI 2-sided [-70.03 to -28.19], Standard Error of Mean 10.529
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Induration: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0023, Mixed Models Analysis; LS mean difference = -29.71, 95% CI 2-sided [-48.52 to -10.89], Standard Error of Mean 9.470
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Scaling: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0009, Mixed Models Analysis; LS mean difference = -36.78, 95% CI 2-sided [-58.08 to -15.49], Standard Error of Mean 10.720
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Erythema: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.5048, Mixed Models Analysis; LS mean difference = 7.03, 95% CI 2-sided [-13.84 to 27.90], Standard Error of Mean 10.495
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Induration: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.4575, Mixed Models Analysis; LS mean difference = 9.16, 95% CI 2-sided [-15.24 to 33.57], Standard Error of Mean 12.273
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Scaling: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.9523, Mixed Models Analysis; LS mean difference = 0.69, 95% CI 2-sided [-22.26 to 23.65], Standard Error of Mean 11.539

19. Secondary Outcome: Percent Change From Baseline in BSA at Month 1, 3 and 6 for Participants With Baseline BSA >0%
Description: Assessment of BSA with psoriasis was performed separately for four body regions: head and neck, upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). The BSA with psoriasis (%) was the sum of the numbers of the handpoints across the 4 body regions.
Time Frame: Baseline, Month 1, 3 and 6
Population: The unit of Percentage is for percent change from baseline: (change from baseline / baseline value)*100% FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo). Analysis only included participants in FAS with Baseline BSA >0%.
  Here "Number of Participants Analyzed" indicates participants included in the MMRM.
  Here "Number analyzed" signifies participants evaluable for this OM at the specific visit.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 131 | 63
Percentage
  Month 1: number analyzed (Participants) | 124 | 60
  Month 1 | -34.82 (4.781) | -6.13 (6.878)
  Month 3: number analyzed (Participants) | 119 | 60
  Month 3 | -51.91 (6.142) | -5.44 (8.671)
  Month 6: number analyzed (Participants) | 111 | 56
  Month 6 | -67.68 (6.225) | -40.91 (8.792)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0008, Mixed Models Analysis; LS mean difference = -28.69, 95% CI 2-sided [-45.24 to -12.15], Standard Error of Mean 8.386
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -46.47, 95% CI 2-sided [-67.45 to -25.49], Standard Error of Mean 10.632
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.0141, Mixed Models Analysis; LS mean difference = -26.76, 95% CI 2-sided [-48.05 to -5.47], Standard Error of Mean 10.778

20. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Psoriatic Arthritis (PGA-PsA) (VAS) at Month 1, 3 and 6
Description: The blinded investigator or qualified assessor assessed how the participant's overall PsA appeared at the time of the visit. The investigator's response was recorded using a 100 mm VAS (Not active at all to Extremely active).
Time Frame: Baseline, Month 1, 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 65
mm
  Month 1: number analyzed (Participants) | 126 | 62
  Month 1 | -17.94 (1.376) | -7.19 (1.965)
  Month 3: number analyzed (Participants) | 122 | 60
  Month 3 | -30.29 (1.479) | -10.84 (2.108)
  Month 6: number analyzed (Participants) | 114 | 56
  Month 6 | -38.75 (1.315) | -32.05 (1.873)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -10.75, 95% CI 2-sided [-15.48 to -6.02], Standard Error of Mean 2.399
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -19.45, 95% CI 2-sided [-24.52 to -14.37], Standard Error of Mean 2.575
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.0039, Mixed Models Analysis; LS mean difference = -6.70, 95% CI 2-sided [-11.22 to -2.18], Standard Error of Mean 2.289

21. Secondary Outcome: Resolution Rate of Dactylitis at Month 1, 3 and 6 for Participants With Baseline Dactylitis Severity Score (DSS) >0
Description: Dactylitis was characterized by swelling of the entire finger or toe. The DSS was a function of finger circumference and tenderness, assessed and summed across all dactylitis digits.
  Resolution rate of dactylitis was defined as achieving DSS =0. Rate was measured in terms of percentage of participants with resolution of dactylitis.
  Dactylitis severity was scored based upon digit tenderness using a scale of 0-3, where 0 = no tenderness and 3 = extreme tenderness, in each digit of the hands and feet. DSS was the sum of the severity of the 20 evaluated digits. The range of total dactylitis scores for a participant would be 0-60 (with a higher score indicating more severe dactylitis).
Time Frame: Month 1, 3 and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline DSS >0. MR was considered to be NR (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 93 | 41
Percentage of participants
  Month 1 | 21.51 | 7.32
  Month 3 | 45.16 | 19.51
  Month 6 | 64.52 | 41.46
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0160, Normal approximation; Difference in percentage of participants = 14.19, 95% CI 2-sided [2.64 to 25.73], Standard Error of Mean 5.89
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.0015, Normal approximation; Difference in percentage of participants = 25.65, 95% CI 2-sided [9.86 to 41.44], Standard Error of Mean 8.06
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.0118, Normal approximation; Difference in percentage of participants = 23.05, 95% CI 2-sided [5.11 to 41.00], Standard Error of Mean 9.16

22. Secondary Outcome: Change From Baseline in DSS for Participant With Baseline DSS >0 at Month 1, 3 and 6
Description: Dactylitis was characterized by swelling of the entire finger or toe. The DSS was a function of finger circumference and tenderness, assessed and summed across all dactylitis digits.
  Dactylitis severity was scored based upon digit tenderness using a scale of 0-3, where 0 = no tenderness and 3 = extreme tenderness, in each digit of the hands and feet. DSS was the sum of the severity of the 20 evaluated digits. The range of total dactylitis scores for a participant would be 0-60 (with a higher score indicating more severe dactylitis).
Time Frame: Baseline, Month 1, 3 and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline DSS >0. Here "Number of Participants Analyzed" indicates participants included in the MMRM.
  Here "Number analyzed" signifies participants evaluable for this OM at the specific visit.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 91 | 40
Unit on a scale
  Month 1: number analyzed (Participants) | 88 | 38
  Month 1 | -4.26 (0.691) | -1.17 (1.052)
  Month 3: number analyzed (Participants) | 86 | 37
  Month 3 | -6.55 (0.543) | -2.49 (0.826)
  Month 6: number analyzed (Participants) | 79 | 34
  Month 6 | -7.80 (0.190) | -6.83 (0.289)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0156, Mixed Models Analysis; LS mean difference = -3.09, 95% CI 2-sided [-5.58 to -0.60], Standard Error of Mean 1.259
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -4.06, 95% CI 2-sided [-6.02 to -2.10], Standard Error of Mean 0.989
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.0061, Mixed Models Analysis; LS mean difference = -0.97, 95% CI 2-sided [-1.65 to -0.28], Standard Error of Mean 0.346

23. Secondary Outcome: Resolution Rate of Enthesitis at Month 1, 3 and 6 for Participants With Baseline Leeds Enthesitis Index (LEI) >0
Description: Resolution rate of enthesitis was defined as percentage of participants achieving enthesitis score (using LEI) =0.
  Rate was measured in terms of percentage of participants with resolution of enthesitis.
  Enthesitis score based upon presence/absence of enthesitis at 6 sites using LEI. Six sites, including (right and left): lateral epicondyle humerus, medial femoral condyle and Achilles tendon insertion, were assessed for enthesitis. LEI was the number of sites with presence of enthesitis.
Time Frame: Month 1, 3 and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline LEI >0. MR was considered to be NR (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 71 | 28
Percentage of participants
  Month 1 | 38.03 | 25.00
  Month 3 | 49.30 | 25.00
  Month 6 | 64.79 | 60.71
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.1930, Normal approximation; Difference in percentage of participants = 13.03, 95% CI 2-sided [-6.59 to 32.64], Standard Error of Mean 10.01
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.0162, Normal approximation; Difference in percentage of participants = 24.30, 95% CI 2-sided [4.48 to 44.11], Standard Error of Mean 10.11
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.7068, Normal approximation; Difference in percentage of participants = 4.07, 95% CI 2-sided [-17.15 to 25.30], Standard Error of Mean 10.83

24. Secondary Outcome: Change From Baseline in LEI for Participant With Baseline LEI >0 at Month 1, 3 and 6
Description: Enthesitis score based upon presence/absence of enthesitis at 6 sites using LEI. Six sites, including (right and left): lateral epicondyle humerus, medial femoral condyle and Achilles tendon insertion, were assessed for enthesitis. LEI was the number of sites with presence of enthesitis.
Time Frame: Baseline, Month 1, 3 and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline LEI >0. Here "Number of Participants Analyzed" indicates participants included in the MMRM.
  Here "Number analyzed" signifies participants evaluable for this OM at the specific visit.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 69 | 27
Unit on a scale
  Month 1: number analyzed (Participants) | 67 | 25
  Month 1 | -1.04 (0.142) | -0.74 (0.231)
  Month 3: number analyzed (Participants) | 63 | 24
  Month 3 | -1.36 (0.155) | -0.99 (0.251)
  Month 6: number analyzed (Participants) | 59 | 23
  Month 6 | -1.87 (0.127) | -1.61 (0.203)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.2811, Mixed Models Analysis; LS mean difference = -0.29, 95% CI 2-sided [-0.83 to 0.25], Standard Error of Mean 0.271
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.2140, Mixed Models Analysis; LS mean difference = -0.37, 95% CI 2-sided [-0.96 to 0.22], Standard Error of Mean 0.295
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.2817, Mixed Models Analysis; LS mean difference = -0.26, 95% CI 2-sided [-0.74 to 0.22], Standard Error of Mean 0.239

25. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score at Month 1, 3 and 6 for Participants With Baseline NAPSI >0
Description: A target finger nail was evaluated using NAPSI scale. Each quadrant of the target nail was graded for nail matrix psoriasis and nail bed psoriasis, giving that 1 target nail a score of 0-8. At the baseline visit, the worst case fingernail was chosen and the same nail evaluated consistently through the entire study.
Time Frame: Baseline, Month 1, 3 and 6
Population: FAS: included all participants randomized and who have received at least one dose of randomized study drug (tofacitinib or placebo).
  Analysis only included participants in FAS with Baseline NAPSI >0. Here "Number of Participants Analyzed" indicates participants included in the MMRM.
  Here "Number analyzed" signifies participants evaluable for this OM at the specific visit.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 96 | 53
Unit on a scale
  Month 1: number analyzed (Participants) | 91 | 50
  Month 1 | -0.26 (0.108) | -0.25 (0.146)
  Month 3: number analyzed (Participants) | 86 | 48
  Month 3 | -1.03 (0.175) | -0.80 (0.235)
  Month 6: number analyzed (Participants) | 82 | 47
  Month 6 | -2.43 (0.189) | -2.10 (0.251)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.9407, Mixed Models Analysis; LS mean difference = -0.01, 95% CI 2-sided [-0.37 to 0.35], Standard Error of Mean 0.182
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.4295, Mixed Models Analysis; LS mean difference = -0.23, 95% CI 2-sided [-0.81 to 0.35], Standard Error of Mean 0.293
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.2946, Mixed Models Analysis; LS mean difference = -0.33, 95% CI 2-sided [-0.95 to 0.29], Standard Error of Mean 0.314

26. Secondary Outcome: Percentage of Participants Achieving Psoriatic Arthritis Response Criteria (PsARC) at Week 2, Month 1, 2, 3, 4, and 6
Description: The PsARC consisted of 4 measurements: Tender Joint Count (68), Swollen Joint Count (66), Physician's Global Assessment of Arthritis (VAS) (0-100 mm), Patient's Global Assessment of Arthritis (VAS) (0-100 mm). In order to be a 'PsARC responder', participant must achieve improvement in 2 of 4 measures, one of which must be joint pain or swelling, without worsening in any measure.
Time Frame: Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 136 | 68
Percentage of participants
  Week 2 | 33.09 | 11.76
  Month 1 | 56.62 | 20.59
  Month 2 | 65.44 | 13.24
  Month 3 | 69.12 | 29.41
  Month 4 | 69.85 | 51.47
  Month 6 | 79.41 | 63.24
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0001, Normal approximation; Difference in percentage of participants = 21.32, 95% CI 2-sided [10.32 to 32.33], Standard Error of Mean 5.62
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 36.03, 95% CI 2-sided [23.31 to 48.75], Standard Error of Mean 6.49
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 52.21, 95% CI 2-sided [40.86 to 63.55], Standard Error of Mean 5.79
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p < 0.0001, Normal approximation; Difference in percentage of participants = 39.71, 95% CI 2-sided [26.38 to 53.03], Standard Error of Mean 6.80
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.0110, Normal approximation; Difference in percentage of participants = 18.38, 95% CI 2-sided [4.22 to 32.55], Standard Error of Mean 7.23
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.0173, Normal approximation; Difference in percentage of participants = 16.18, 95% CI 2-sided [2.85 to 29.50], Standard Error of Mean 6.80

27. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS)28-3 (CRP) at Week 2, Month 1, 2, 3, 4, and 6
Description: The DAS was a derived measurement with differential weighting given to each component. The components of the DAS 28-3 arthritis assessment were: Tender/Painful Joint Count (28), Swollen Joint Count (28), CRP (refer to above OMs for more details of these components). DAS28 scores range from 0 to 9.4. A DAS28-3 (CRP) score higher than 5.1 indicates high disease activity, a DAS28-3 (CRP) score less than 3.2 indicates low disease activity, and a DAS28-3 (CRP) score less than 2.6 indicates clinical remission. A higher score represented a more severe disease activity, and a negative change from baseline indicates improvement.
  DAS28-3(CRP)=[0.56*sqrt(TJC28)+0.28*sqrt(SJC28)+0.36*ln(CRP+1)]*1.10+1.15, where sqrt() refers to the square root, and ln() refers to the natural logarithm.
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4, and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 135 | 67
Unit on a scale
  Week 2: number analyzed (Participants) | 131 | 66
  Week 2 | -0.68 (0.046) | -0.05 (0.065)
  Month 1: number analyzed (Participants) | 126 | 62
  Month 1 | -0.92 (0.054) | -0.12 (0.077)
  Month 2: number analyzed (Participants) | 117 | 58
  Month 2 | -1.13 (0.060) | -0.26 (0.086)
  Month 3: number analyzed (Participants) | 123 | 60
  Month 3 | -1.34 (0.070) | -0.30 (0.100)
  Month 4: number analyzed (Participants) | 115 | 57
  Month 4 | -1.59 (0.074) | -1.16 (0.105)
  Month 6: number analyzed (Participants) | 115 | 56
  Month 6 | -1.85 (0.083) | -1.63 (0.119)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.63, 95% CI 2-sided [-0.79 to -0.47], Standard Error of Mean 0.080
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.81, 95% CI 2-sided [-0.99 to -0.62], Standard Error of Mean 0.095
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.87, 95% CI 2-sided [-1.08 to -0.66], Standard Error of Mean 0.105
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.04, 95% CI 2-sided [-1.28 to -0.80], Standard Error of Mean 0.122
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0009, Mixed Models Analysis; LS mean difference = -0.44, 95% CI 2-sided [-0.69 to -0.18], Standard Error of Mean 0.129
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.1202, Mixed Models Analysis; LS mean difference = -0.23, 95% CI 2-sided [-0.51 to 0.06], Standard Error of Mean 0.145

28. Secondary Outcome: Change From Baseline in Short-Form-36 Health Survey (SF-36) Version 2, Acute at Month 1, 3 and 6
Description: The SF 36 v.2 (Acute) was a 36 item generic health status measure. It measured 8 general health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. These domains were summarized as physical and mental component summary scores. The score range for the physical and mental health scores was 0-100 (100=highest level of functioning).
Time Frame: Baseline, Month 1, 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 65
Unit on a scale
  Month 1: Physical Functioning Domain: number analyzed (Participants) | 132 | 64
  Month 1: Physical Functioning Domain | 3.53 (0.570) | -0.19 (0.819)
  Month 1: Role-Physical Domain: number analyzed (Participants) | 132 | 64
  Month 1: Role-Physical Domain | 3.93 (0.630) | 0.75 (0.903)
  Month 1: Bodily Pain Domain: number analyzed (Participants) | 132 | 64
  Month 1: Bodily Pain Domain | 5.58 (0.492) | 2.47 (0.706)
  Month 1: General Health Domain: number analyzed (Participants) | 132 | 54
  Month 1: General Health Domain | 3.33 (0.537) | -0.21 (0.770)
  Month 1: Vitality Domain: number analyzed (Participants) | 132 | 64
  Month 1: Vitality Domain | 3.12 (0.687) | 0.08 (0.987)
  Month 1: Social Function Domain: number analyzed (Participants) | 132 | 64
  Month 1: Social Function Domain | 2.65 (0.637) | 0.07 (0.915)
  Month 1: Role-Emotional Domain: number analyzed (Participants) | 132 | 64
  Month 1: Role-Emotional Domain | 3.19 (0.763) | 1.15 (1.095)
  Month 1: Mental Health Domain: number analyzed (Participants) | 132 | 64
  Month 1: Mental Health Domain | 1.77 (0.669) | -0.14 (0.960)
  Month 1: Physical Component Summary: number analyzed (Participants) | 132 | 64
  Month 1: Physical Component Summary | 4.52 (0.437) | 0.76 (0.626)
  Month 1: Mental Component Summary: number analyzed (Participants) | 132 | 64
  Month 1: Mental Component Summary | 1.85 (0.671) | 0.07 (0.964)
  Month 3: Physical Functioning Domain: number analyzed (Participants) | 125 | 62
  Month 3: Physical Functioning Domain | 4.33 (0.705) | 1.80 (1.001)
  Month 3: Role-Physical Domain: number analyzed (Participants) | 125 | 62
  Month 3: Role-Physical Domain | 5.94 (0.705) | 1.52 (1.004)
  Month 3: Bodily Pain Domain: number analyzed (Participants) | 125 | 62
  Month 3: Bodily Pain Domain | 7.60 (0.614) | 2.30 (0.874)
  Month 3: General Health Domain: number analyzed (Participants) | 125 | 62
  Month 3: General Health Domain | 5.11 (0.725) | -0.16 (1.032)
  Month 3: Vitality Domain: number analyzed (Participants) | 125 | 62
  Month 3: Vitality Domain | 3.81 (0.784) | 1.71 (1.116)
  Month 3: Social Function Domain: number analyzed (Participants) | 125 | 62
  Month 3: Social Function Domain | 4.75 (0.681) | 0.42 (0.969)
  Month 3: Role-Emotional Domain: number analyzed (Participants) | 125 | 62
  Month 3: Role-Emotional Domain | 5.30 (0.795) | 1.86 (1.132)
  Month 3: Mental Health Domain: number analyzed (Participants) | 125 | 62
  Month 3: Mental Health Domain | 2.90 (0.728) | -0.58 (1.036)
  Month 3: Physical Component Summary: number analyzed (Participants) | 125 | 62
  Month 3: Physical Component Summary | 6.02 (0.567) | 1.85 (0.806)
  Month 3: Mental Component Summary: number analyzed (Participants) | 125 | 62
  Month 3: Mental Component Summary | 3.38 (0.715) | 0.11 (1.019)
  Month 6: Physical Functioning Domain: number analyzed (Participants) | 126 | 61
  Month 6: Physical Functioning Domain | 6.35 (0.600) | 5.96 (0.860)
  Month 6: Role-Physical Domain: number analyzed (Participants) | 126 | 61
  Month 6: Role-Physical Domain | 6.88 (0.705) | 5.84 (1.011)
  Month 6: Bodily Pain Domain: number analyzed (Participants) | 126 | 61
  Month 6: Bodily Pain Domain | 10.68 (0.678) | 10.31 (0.973)
  Month 6: General Health Domain: number analyzed (Participants) | 126 | 61
  Month 6: General Health Domain | 5.54 (0.762) | 4.32 (1.091)
  Month 6: Vitality Domain: number analyzed (Participants) | 126 | 61
  Month 6: Vitality Domain | 5.60 (0.868) | 3.61 (1.246)
  Month 6: Social Function Domain: number analyzed (Participants) | 126 | 61
  Month 6: Social Function Domain | 5.58 (0.691) | 5.30 (0.991)
  Month 6: Role-Emotional Domain: number analyzed (Participants) | 126 | 61
  Month 6: Role-Emotional Domain | 6.35 (0.782) | 4.12 (1.121)
  Month 6: Mental Health Domain: number analyzed (Participants) | 126 | 61
  Month 6: Mental Health Domain | 3.68 (0.795) | 2.97 (1.141)
  Month 6: Physical Component Summary: number analyzed (Participants) | 126 | 61
  Month 6: Physical Component Summary | 7.94 (0.580) | 7.55 (0.831)
  Month 6: Mental Component Summary: number analyzed (Participants) | 126 | 61
  Month 6: Mental Component Summary | 3.99 (0.812) | 2.20 (1.166)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Physical Functioning Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0003, Mixed Models Analysis; LS mean difference = 3.72, 95% CI 2-sided [1.76 to 5.69], Standard Error of Mean 0.998
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Role - Physical Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0043, Mixed Models Analysis; LS mean difference = 3.18, 95% CI 2-sided [1.01 to 5.35], Standard Error of Mean 1.102
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Bodily Pain Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0004, Mixed Models Analysis; LS mean difference = 3.12, 95% CI 2-sided [1.42 to 4.82], Standard Error of Mean 0.861
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, General Health Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS mean difference = 3.54, 95% CI 2-sided [1.69 to 5.39], Standard Error of Mean 0.938
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Vitality Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0123, Mixed Models Analysis; LS mean difference = 3.04, 95% CI 2-sided [0.67 to 5.41], Standard Error of Mean 1.203
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Social Function Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0216, Mixed Models Analysis; LS mean difference = 2.58, 95% CI 2-sided [0.38 to 4.78], Standard Error of Mean 1.115
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Role - Emotional Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1290, Mixed Models Analysis; LS mean difference = 2.04, 95% CI 2-sided [-0.60 to 4.67], Standard Error of Mean 1.336
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Mental Health Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1043, Mixed Models Analysis; LS mean difference = 1.91, 95% CI 2-sided [-0.40 to 4.22], Standard Error of Mean 1.172
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Physical Component Summary: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 3.77, 95% CI 2-sided [2.26 to 5.27], Standard Error of Mean 0.763
Statistical Analysis 10: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Mental Component Summary: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1318, Mixed Models Analysis; LS mean difference = 1.78, 95% CI 2-sided [-0.54 to 4.10], Standard Error of Mean 1.178
Statistical Analysis 11: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Physical Functioning Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0402, Mixed Models Analysis; LS mean difference = 2.53, 95% CI 2-sided [0.11 to 4.95], Standard Error of Mean 1.225
Statistical Analysis 12: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Role - Physical Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0004, Mixed Models Analysis; LS mean difference = 4.41, 95% CI 2-sided [1.99 to 6.83], Standard Error of Mean 1.227
Statistical Analysis 13: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Bodily Pain Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 5.29, 95% CI 2-sided [3.18 to 7.40], Standard Error of Mean 1.069
Statistical Analysis 14: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, General Health Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 5.28, 95% CI 2-sided [2.79 to 7.76], Standard Error of Mean 1.261
Statistical Analysis 15: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Vitality Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1254, Mixed Models Analysis; LS mean difference = 2.10, 95% CI 2-sided [-0.59 to 4.80], Standard Error of Mean 1.366
Statistical Analysis 16: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Social Function Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0003, Mixed Models Analysis; LS mean difference = 4.34, 95% CI 2-sided [2.00 to 6.68], Standard Error of Mean 1.186
Statistical Analysis 17: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Role - Emotional Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0140, Mixed Models Analysis; LS mean difference = 3.43, 95% CI 2-sided [0.70 to 6.16], Standard Error of Mean 1.384
Statistical Analysis 18: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Mental Health Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0067, Mixed Models Analysis; LS mean difference = 3.47, 95% CI 2-sided [0.97 to 5.98], Standard Error of Mean 1.268
Statistical Analysis 19: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Physical Component Summary: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 4.17, 95% CI 2-sided [2.23 to 6.12], Standard Error of Mean 0.986
Statistical Analysis 20: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Mental Component Summary: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0094, Mixed Models Analysis; LS mean difference = 3.27, 95% CI 2-sided [0.81 to 5.73], Standard Error of Mean 1.248
Statistical Analysis 21: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Physical Functioning Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.7098, Mixed Models Analysis; LS mean difference = 0.39, 95% CI 2-sided [-1.68 to 2.46], Standard Error of Mean 1.049
Statistical Analysis 22: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Role - Physical Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.4019, Mixed Models Analysis; LS mean difference = 1.04, 95% CI 2-sided [-1.40 to 3.47], Standard Error of Mean 1.234
Statistical Analysis 23: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Bodily Pain Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.7537, Mixed Models Analysis; LS mean difference = 0.37, 95% CI 2-sided [-1.97 to 2.71], Standard Error of Mean 1.186
Statistical Analysis 24: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, General Health Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.3595, Mixed Models Analysis; LS mean difference = 1.22, 95% CI 2-sided [-1.40 to 3.85], Standard Error of Mean 1.330
Statistical Analysis 25: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Vitality Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1919, Mixed Models Analysis; LS mean difference = 1.99, 95% CI 2-sided [-1.01 to 4.99], Standard Error of Mean 1.520
Statistical Analysis 26: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Social Function Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.8163, Mixed Models Analysis; LS mean difference = 0.28, 95% CI 2-sided [-2.10 to 2.67], Standard Error of Mean 1.209
Statistical Analysis 27: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Role - Emotional Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1048, Mixed Models Analysis; LS mean difference = 2.23, 95% CI 2-sided [-0.47 to 4.93], Standard Error of Mean 1.368
Statistical Analysis 28: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Mental Health Domain: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.6118, Mixed Models Analysis; LS mean difference = 0.71, 95% CI 2-sided [-2.04 to 3.45], Standard Error of Mean 1.392
Statistical Analysis 29: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Physical Component Summary: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.6996, Mixed Models Analysis; LS mean difference = 0.39, 95% CI 2-sided [-1.61 to 2.39], Standard Error of Mean 1.014
Statistical Analysis 30: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Mental Component Summary: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.2122, Mixed Models Analysis; LS mean difference = 1.78, 95% CI 2-sided [-1.03 to 4.59], Standard Error of Mean 1.424

29. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions 3 Levels (EQ-5D-3L) Domain Scores at Month 1, 3 and 6
Description: On the EQ-5D (participant version, 3 categories of response per question), 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) were assessed. The status of each dimension had three possible responses with the corresponding scores of 1 (no problem), 2 (some problems) and 3 (severe problems).
Time Frame: Baseline, Month 1, 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 65
Unit on a scale
  Month 1: Mobility: number analyzed (Participants) | 132 | 64
  Month 1: Mobility | -0.14 (0.038) | -0.02 (0.055)
  Month 1: Self-Care: number analyzed (Participants) | 132 | 64
  Month 1: Self-Care | -0.15 (0.031) | 0.01 (0.045)
  Month 1: Usual Activities: number analyzed (Participants) | 132 | 64
  Month 1: Usual Activities | -0.19 (0.039) | -0.05 (0.056)
  Month 1: Pain/Discomfort: number analyzed (Participants) | 132 | 54
  Month 1: Pain/Discomfort | -0.28 (0.037) | -0.15 (0.054)
  Month 1: Anxiety/Depression: number analyzed (Participants) | 132 | 64
  Month 1: Anxiety/Depression | -0.19 (0.036) | -0.11 (0.051)
  Month 3: Mobility: number analyzed (Participants) | 125 | 62
  Month 3: Mobility | -0.24 (0.037) | 0.01 (0.053)
  Month 3: Self-Care: number analyzed (Participants) | 125 | 62
  Month 3: Self-Care | -0.16 (0.033) | 0.02 (0.047)
  Month 3: Usual Activities: number analyzed (Participants) | 125 | 62
  Month 3: Usual Activities | -0.32 (0.040) | 0.01 (0.057)
  Month 3: Pain/Discomfort: number analyzed (Participants) | 125 | 62
  Month 3: Pain/Discomfort | -0.38 (0.042) | -0.10 (0.059)
  Month 3: Anxiety/Depression: number analyzed (Participants) | 125 | 62
  Month 3: Anxiety/Depression | -0.23 (0.036) | -0.12 (0.052)
  Month 6: Mobility: number analyzed (Participants) | 126 | 61
  Month 6: Mobility | -0.32 (0.032) | -0.22 (0.046)
  Month 6: Self-Care: number analyzed (Participants) | 126 | 61
  Month 6: Self-Care | -0.22 (0.028) | -0.19 (0.040)
  Month 6: Usual Activities: number analyzed (Participants) | 126 | 61
  Month 6: Usual Activities | -0.36 (0.037) | -0.25 (0.053)
  Month 6: Pain/Discomfort: number analyzed (Participants) | 126 | 61
  Month 6: Pain/Discomfort | -0.56 (0.046) | -0.56 (0.065)
  Month 6: Anxiety/Depression: number analyzed (Participants) | 126 | 61
  Month 6: Anxiety/Depression | -0.22 (0.038) | -0.28 (0.055)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Mobility: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0722, Mixed Models Analysis; LS mean difference = -0.12, 95% CI 2-sided [-0.25 to 0.01], Standard Error of Mean 0.067
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Self-Care: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0035, Mixed Models Analysis; LS mean difference = -0.16, 95% CI 2-sided [-0.27 to -0.05], Standard Error of Mean 0.055
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Usual Activities: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0475, Mixed Models Analysis; LS mean difference = -0.14, 95% CI 2-sided [-0.27 to 0.00], Standard Error of Mean 0.069
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Pain/Discomfort: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0537, Mixed Models Analysis; LS mean difference = -0.13, 95% CI 2-sided [-0.26 to 0.00], Standard Error of Mean 0.066
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 1, Anxiety/Depression: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1977, Mixed Models Analysis; LS mean difference = -0.08, 95% CI 2-sided [-0.20 to 0.04], Standard Error of Mean 0.062
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Mobility: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0001, Mixed Models Analysis; LS mean difference = -0.25, 95% CI 2-sided [-0.38 to -0.13], Standard Error of Mean 0.064
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Self-Care: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0018, Mixed Models Analysis; LS mean difference = -0.18, 95% CI 2-sided [-0.29 to -0.07], Standard Error of Mean 0.057
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Usual Activities: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.33, 95% CI 2-sided [-0.47 to -0.19], Standard Error of Mean 0.070
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Pain/Discomfort: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS mean difference = -0.28, 95% CI 2-sided [-0.42 to -0.14], Standard Error of Mean 0.073
Statistical Analysis 10: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Anxiety/Depression: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0835, Mixed Models Analysis; LS mean difference = -0.11, 95% CI 2-sided [-0.23 to 0.01], Standard Error of Mean 0.063
Statistical Analysis 11: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Mobility: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0825, Mixed Models Analysis; LS mean difference = -0.10, 95% CI 2-sided [-0.21 to 0.01], Standard Error of Mean 0.056
Statistical Analysis 12: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Self-Care: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.5616, Mixed Models Analysis; LS mean difference = -0.03, 95% CI 2-sided [-0.13 to 0.07], Standard Error of Mean 0.049
Statistical Analysis 13: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Usual Activities: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.0748, Mixed Models Analysis; LS mean difference = -0.12, 95% CI 2-sided [-0.24 to 0.01], Standard Error of Mean 0.065
Statistical Analysis 14: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Pain/Discomfort: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.9477, Mixed Models Analysis; LS mean difference = 0.01, 95% CI 2-sided [-0.15 to 0.16], Standard Error of Mean 0.080
Statistical Analysis 15: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Anxiety/Depression: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.3829, Mixed Models Analysis; LS mean difference = 0.06, 95% CI 2-sided [-0.07 to 0.19], Standard Error of Mean 0.067

30. Secondary Outcome: Change From Baseline in EuroQol Visual Analogue Scale (EQ-VAS) Score at Month 1, 3 and 6
Description: The EQ-VAS recorded the patient's self-rated health on a vertical visual analogue scale where the endpoint was labelled 'Best imaginable health state' and 'Worst imaginable health state'. Based on the patient's mark on the VAS form a score ranging from 0 to 100 mm was recorded.
Time Frame: Baseline, Month 1, 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 65
mm
  Month 1: number analyzed (Participants) | 132 | 64
  Month 1 | 9.88 (1.191) | 3.87 (1.710)
  Month 3: number analyzed (Participants) | 125 | 62
  Month 3 | 12.48 (1.484) | 1.68 (2.108)
  Month 6: number analyzed (Participants) | 126 | 61
  Month 6 | 18.52 (1.398) | 17.60 (2.002)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0044, Mixed Models Analysis; LS mean difference = 6.01, 95% CI 2-sided [1.90 to 10.12], Standard Error of Mean 2.084
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 10.80, 95% CI 2-sided [5.71 to 15.88], Standard Error of Mean 2.578
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.7062, Mixed Models Analysis; LS mean difference = 0.92, 95% CI 2-sided [-3.90 to 5.74], Standard Error of Mean 2.442

31. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment-Psoriatic Arthritis (WPAI-PsA) at Month 3 and 6: Work Time Missed, Impairment While Working, Overall Work Impairment
Description: The WPAI-PsA was a 6-item questionnaire that measured absenteeism (work time missed), presenteesism (impairment at work/reduced on -the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism) and activity impairment. WPAI-PsA outcomes were expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Month 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 63 | 34
Percentage
  Month 3: Work Time Missed: number analyzed (Participants) | 59 | 32
  Month 3: Work Time Missed | -1.01 (1.422) | -1.86 (1.933)
  Month 3: Impairment While Working: number analyzed (Participants) | 59 | 32
  Month 3: Impairment While Working | -16.11 (2.703) | -9.77 (3.673)
  Month 3: Overall Work Impairment: number analyzed (Participants) | 59 | 32
  Month 3: Overall Work Impairment | -16.67 (2.789) | -10.45 (3.790)
  Month 6: Work Time Missed: number analyzed (Participants) | 56 | 26
  Month 6: Work Time Missed | -1.09 (1.451) | -0.01 (2.132)
  Month 6: Impairment While Working: number analyzed (Participants) | 56 | 27
  Month 6: Impairment While Working | -21.11 (2.819) | -18.73 (4.014)
  Month 6: Overall Work Impairment: number analyzed (Participants) | 56 | 26
  Month 6: Overall Work Impairment | -20.91 (3.031) | -18.28 (4.389)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Work Time Missed: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.7228, Mixed Models Analysis; LS mean difference = 0.86, 95% CI 2-sided [-3.92 to 5.63], Standard Error of Mean 2.404
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Impairment While Working: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1682, Mixed Models Analysis; LS mean difference = -6.34, 95% CI 2-sided [-15.39 to 2.72], Standard Error of Mean 4.561
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Overall Work Impairment: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.1900, Mixed Models Analysis; LS mean difference = -6.21, 95% CI 2-sided [-15.56 to 3.13], Standard Error of Mean 4.707
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Work Time Missed: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.6757, Mixed Models Analysis; LS mean difference = -1.08, 95% CI 2-sided [-6.22 to 4.05], Standard Error of Mean 2.581
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Impairment While Working: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.6285, Mixed Models Analysis; LS mean difference = -2.38, 95% CI 2-sided [-12.13 to 7.37], Standard Error of Mean 4.905
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Overall Work Impairment: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.6228, Mixed Models Analysis; LS mean difference = -2.63, 95% CI 2-sided [-13.23 to 7.97], Standard Error of Mean 5.333

32. Secondary Outcome: Change From Baseline in WPAI-PsA at Month 3 and 6: Activity Impairment
Description: The WPAI-PsA was a 6-item questionnaire that measured absenteeism (work time missed), presenteesism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism) and activity impairment. WPAI-PsA outcomes were expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Month 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 129 | 64
Percentage
  Month 3: Activity Impairment: number analyzed (Participants) | 125 | 62
  Month 3: Activity Impairment | -17.20 (1.778) | -4.39 (2.525)
  Month 6: Activity Impairment: number analyzed (Participants) | 126 | 61
  Month 6: Activity Impairment | -21.91 (1.805) | -22.97 (2.589)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 3, Activity Impairment: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -12.81, 95% CI 2-sided [-18.90 to -6.72], Standard Error of Mean 3.089
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Month 6, Activity Impairment: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, and baseline value; Test type: Superiority; p = 0.7384, Mixed Models Analysis; LS mean difference = 1.06, 95% CI 2-sided [-5.17 to 7.28], Standard Error of Mean 3.157

ADVERSE EVENTS:
Time Frame: For "Tofacitinib: Up to Month 3" arm and "Placebo: Up to Month 3" arm: From the baseline to Month 3. For "Tofacitinib: Up to Month 6" arm and "Placebo Then Tofacitinib: Up to Month 6" arm: From the baseline to up to 42 days after the last dose of the study treatment (up to 7.5 months).
Description: Same event may appear as AE and serious AE. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who were randomized and received at least one dose of the investigational product (i.e., tofacitinib or placebo).
Groups:
- Tofacitinib: Up to Month 3: Participants received Tofacitinib 5 mg tablets BID for 3 months.
- Placebo: Up to Month 3: Participants received tofacitinib matching placebo tablets BID for 3 months
- Tofacitinib: Up to Month 6: Participants received tofacitinib 5 mg tablets twice daily for 6 months.
- Placebo Then Tofacitinib: Up to Month 6: Participants received tofacitinib matching placebo tablets BID for 3 months, followed by tofacitinib tablets 5 mg BID for next 3 months.
Arm/Group | Tofacitinib: Up to Month 3 | Placebo: Up to Month 3 | Tofacitinib: Up to Month 6 | Placebo Then Tofacitinib: Up to Month 6
All-Cause Mortality (participants affected / at risk) | 0/136 | 1/68 | 0/136 | 1/68
Serious Adverse Events (participants affected / at risk) | 0/136 | 3/68 | 2/136 | 5/68
Other Adverse Events (participants affected / at risk) | 60/136 | 16/68 | 94/136 | 37/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib: Up to Month 3 (N=136) | Placebo: Up to Month 3 (N=68) | Tofacitinib: Up to Month 6 (N=136) | Placebo Then Tofacitinib: Up to Month 6 (N=68)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib: Up to Month 3 (N=136) | Placebo: Up to Month 3 (N=68) | Tofacitinib: Up to Month 6 (N=136) | Placebo Then Tofacitinib: Up to Month 6 (N=68)
Abdominal discomfort (Gastrointestinal disorders) | 9 (13) | 1 (1) | 9 (16) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 2 (2) | 12 (16) | 2 (4)
Upper respiratory tract infection (Infections and infestations) | 25 (27) | 7 (9) | 36 (45) | 7 (9)
Alanine aminotransferase increased (Investigations) | 7 (7) | 4 (4) | 11 (12) | 5 (7)
Blood creatine phosphokinase increased (Investigations) | 9 (10) | 1 (1) | 20 (21) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (9) | 2 (2) | 14 (15) | 6 (8)
Dizziness (Nervous system disorders) | 7 (8) | 1 (1) | 7 (8) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 12 (12) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 11 (11) | 4 (5)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 5 (7) | 4 (5)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 8 (9) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 9 (15) | 3 (3)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT03486457/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03486457/SAP_001.pdf